CLINICAL TRIAL: NCT02388893
Title: Endocarditis Registry of the University Hospital of Cologne (ER-UHC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Guido Michels, Dr. Guido Michels, University of Cologne
Other Study IDs: 14-221; 14-221 (Other: Ethics committee of the University of Cologne)
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
As recommended in the Guidelines on the prevention, diagnosis, and treatment of infective endocarditis (IE) patients with IE should be evaluated and managed by a multispecialty team including an cardiologist, infectious disease specialist, and cardiac surgeon. Our registry is a prospective, national registry of patients with IE. From January 2013 data from endocarditis board were prospectively recorded using standard definitions during the hospitalization. Patient demographics, clinical, laboratory, and imaging data at the time of IE diagnosis, as well as treatment outcomes were entered into the ER-UHC database.

DETAILED DESCRIPTION:
The primary endpoint will be the 1 year all-cause mortality after treatment begins of IE. We will use 1 year all-cause mortality as the primary endpoint because it has been demonstrated that a period of at least 6 months is necessary to offset the early postoperative mortality related to valve surgery. We also looked at all-cause in-hospital mortality as a secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* All patients with patients with definitive infective endocarditis

Exclusion Criteria:

* childs

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with definitive IE
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 1 year
  1-year all-cause mortality

SECONDARY OUTCOMES:
Inhospital all-cause mortality | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Guido Michels, Prof. Dr., Principal Investigator — Heart Center, University of Cologne, Germany
Locations (1):
- Heart Center of the University of Cologne, Cologne, Germany